CLINICAL TRIAL: NCT03915704
Title: Effects of Two Different Methods During Intramuscular Injections On Pain, Fear, and Satisfaction in Pediatric Emergency Department Patients: A Randomized Controlled Trial
Brief Title: Intramuscular Injection-Related Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Burcu Aykanat Girgin, PhD RN, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07112018139
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pain; Fear
Keywords: pain management; intramuscular injection; non-pharmacological method
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy (Experimental): Buzzy was placed 3-5 cm above the injection site 60 sec before the injection and used until the procedure was completed. The Buzzy application to all children in this group was done by the second researcher. After the injection, the ice pack was wiped with 70% alcohol and frozen again by freezing.
  Interventions: Device: Buzzy
- Shotblocker (Experimental): ShotBlocker is a small, flat, yellow horseshoe-shaped plastic tool that is non-invasive, appropriate for every age group, does not have the characteristics of medication or adverse effects. ShotBlocker has short, blunt points that provide contact with skin on one side, and a hole that exposes the injection site in the middle of the tool. It is used by being held on the skin surface during injection. The pointed surface of the tool is placed on the administration area right before the injection
  Interventions: Device: Shotblocker
- Control (Experimental): No intervention was performed to reduce pain and fear in the control group.
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Shotblocker — Injection was administered with ShotBlocker.The Shotblocker application to all children in this group was done by the second researcher. After the injection, the shotblocker was wiped with 70% alcohol.
  Arms: Shotblocker
Procedure: Control — No intervention was made in the children.
  Arms: Control
Device: Buzzy — Buzzy was placed 3-5 cm above the injection site 60 sec before the injection and used until the procedure was completed.The Buzzy application to all children in this group was done by the second researcher. After the injection, the ice pack was wiped with 70% alcohol and frozen again by freezing.
  Arms: Buzzy

SUMMARY:
The study is an experimental randomized controlled study conducted to compare the effect of buzzy and shotblocker methods applied during intramuscular injection from on pain and fear level in 6-12 year-old children. The sample of the study consisted of 90 children aged between 6 and 12 years who were diagnosed with upper and lower tract respiratory infections and received intramuscular injection of ceftriaxone at the pediatric emergency department of a university hospital in İstanbul between November 2018 and April 2019. The children were divided into 3 groups of 30 people, including shotblocker, buzzy, and control groups. Each intervention and control group was matched in terms of gender. In the study, the randomization of the sample group was performed by using stratification and block randomization methods.

DETAILED DESCRIPTION:
The study is a randomized controlled, non-blinded, experimental trial. The sample of the study consisted of 90 children aged between 6 and 12 years who were diagnosed with upper and lower tract respiratory infections and received intramuscular injection of ceftriaxone at the pediatric emergency department of a university hospital in İstanbul between November 2018 and April 2019. The children were recruited into the study on the basis of the following criteria: being aged between 6-12, requiring for ceftriaxone intramuscular injection because of upper and lower respiratory tract infections, being cognitively able to rate pain and fear scales, and voluntariliy signing the written informed consent. Children were excluded if they had a disease causing chronic pain, received analgesics within the last 6 hours, with pacemakers, had infection, rash, or detoriorated skin integrity in the site where the injection was to be made, had nerve damage in the injection site, had critical or unstable health status, had intellectual disability, reynaud's syndrome, and sickle cell disease, and were unwilling to participate in the study. Also, the parents were eligible for the participation when meeting the following inclusion criteria: 1) be healthy in terms of neurologic functions, 2) communicate verbally, 3) understand and read Turkish, and 4) voluntarily sign the written informed consent. The sample size should be determined as minimum 30 in both experimental and control groups in the experimental studies and parametric measurements. Therefore, 90 children who met the inclusion criteria of the study between specified dates were enrolled and each group included 30 children including two experimental groups and a control group. In order to prevent bias and increase the validity of the data, the pain and fear scores of the children before and after the procedure were assessed by three different groups as children participating in the study (n:90), their parents (n:90), and a researcher specialized in pediatric nursing (n:1).

The children were included in one of the 3 study groups, including buzzy, shotblocker, and control group without any intervention. In order to control the effect of gender on pain, the children were stratified into study groups based on their gender and selected by using block randomization methods in three study groups. The children were randomized to the related study group by drawing one of the study groups in the cloth bags prepared for the girls (pink) and the boys (blue). Papers with the same color and folding pattern representing the four groups (1,2,3,4) were thrown in the bags. In order to provide a randomized distribution and to reduce all negative effects, the children were asked to take randomly a paper from the bag according to the gender after making the necessary explanation to the parents and their children so that the groups became self-balancing. A total of 30 children including 15 girls and 15 boys were included in each group after intervention and control groups were matched in themselves in terms of gender.

The study followed the CONSORT guideline for reporting randomized controlled trials. The pain level of children before and after the injection was assessed using Wong-Baker FACES Pain Rating Scale. To assess the pain level of the children, the children were asked to evaluate themselves, and their parents and first researcher were requested to evaluate the children's pain level immediately before and after the injection. The responses of the children, their parents, and the first researcher were scored blindly. The fear level of children before and after the injection was assessed using Children's Fear Scale. To assess the fear level of the children, the children were asked to evaluate themselves, and their parents and first researcher were requested to evaluate the children's fear level immediately before and after the injection. The responses of the children, their parents, and the first researcher were scored blindly.

ELIGIBILITY:
Inclusion Criteria:

1. being aged between 6-12,
2. requiring for ceftriaxone intramuscular injection because of upper and lower respiratory tract infections,
3. being cognitively able to rate pain and fear scales, and voluntariliy signing the written informed consent.

Exclusion Criteria:

1. having a disease causing chronic pain,
2. receiving analgesics within the last 6 hours, with pacemakers,
3. having infection, rash, or detoriorated skin integrity in the site where the injection was to be made, had nerve damage in the injection site,
4. having critical or unstable health status, had intellectual disability, reynaud's syndrome, and sickle cell disease
5. being unwilling to participate in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Pain severity | 5 Months
  The pain level of children before and after the injection was assessed using Wong-Baker FACES Pain Rating Scale. To assess the pain level of the children, the children were asked to evaluate themselves, and their parents and first researcher were requested to evaluate the children's pain level immediately before and after the injection. The responses of the children, their parents, and the first researcher were scored blindly. This scale has the faces and the pain score is determined according to the numerical values given to the faces. While smiley face "0 point" shows lack of pain, crying face "10 points" refer to severe pain (Merkel & Malviya, 2000). The validity and reliability of this scale was conducted

SECONDARY OUTCOMES:
Fear Levels | 5 Months
  The fear level of children before and after the injection was assessed using Children's Fear Scale. To assess the fear level of the children, the children were asked to evaluate themselves, and their parents and first researcher were requested to evaluate the children's fear level immediately before and after the injection. The responses of the children, their parents, and the first researcher were scored blindly.This scale has five facial expression and the fear is scored according to the numerical values given to the faces on the scale. The leftmost face "0 point" in the scale represents that the child has no fear and the rightmost face "4 points" represent that the child is frightened a lot.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Aykanat Girgin, PhD RN, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)